CLINICAL TRIAL: NCT06936020
Title: Effects of Peripheral Somatosensory Stimulation Via Mechanical Pressure on Lower Limb Muscle Strength in Healthy Subjects.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Facultat de ciencies de la Salut Universitat Ramon Llull (Other)
Responsible Party: Principal Investigator, Pedro Victor López Plaza, Principal Investigator,, Facultat de ciencies de la Salut Universitat Ramon Llull
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-04-08
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: The design of this study is a randomized crossover clinical trial. All participants (n=36) will randomly receive both the Active and Sham proprioceptive stimulation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The control group (CG) (No Intervention): he control group (CG) will have the proprioceptive stimulation device placed on the motor points of the quadriceps muscle without the application of deep sensory stimulation throughout the entire evaluation period of Maximum Strength (MS) via Mean Velocity (MV), including rest periods.
- The Experimental Group 1 (EG1) (Experimental): The Experimental Group 1 (EG1) will have the device placed on the motor points of the quadriceps muscle with deep peripheral sensory stimulation applied via the device's plungers throughout the entire evaluation period of Maximum Strength (MS) via Mean Velocity (MV), including rest periods.
  Interventions: Other: deep peripheral sensory stimulation
- The Experimental Group 2 (EG2) (Experimental): The Experimental Group 2 (EG2) will have the device placed on the motor points of the quadriceps muscle with deep peripheral sensory stimulation applied via the device's plungers, but only during the rest periods between repetitions in the evaluation process of Maximum Strength (MS) via Mean Velocity (MV), applied continuously for 15 seconds at 20-second intervals over a total of 5 minutes.
  Interventions: Other: deep peripheral sensory stimulation

INTERVENTIONS:
Other: deep peripheral sensory stimulation — The proprioceptive stimulus will consist of intermittent mechanical pressure on the skin, localized at the neuromuscular motor points of the rectus femoris, vastus lateralis, and vastus medialis of the quadriceps. The tissue subjected to this precise pressure in areas of high neuromuscular innervation facilitates the stimulation of kinesthetic cortical sensitivity. The experimental group (EG) will be randomly and crosswise subdivided into two groups, so that both receive the intervention in two different modalities at two different times.
  Arms: The Experimental Group 1 (EG1); The Experimental Group 2 (EG2)

SUMMARY:
The proprioceptive system and strength are closely related within the sensorimotor system: proprioception enables effective and coordinated muscle activation (including intramuscular and intermuscular coordination or synergistic abilities), which is essential for maintaining the functional stability of joints and preventing injuries-in short, for controlling motor patterns. This principle provides a window through which changes in strength can be observed via peripheral proprioceptive stimulation that activates the muscular system with the goal of increasing recruitment. This justifies the implementation of proprioceptive input in approaches aimed at motor learning.

DETAILED DESCRIPTION:
Objective: To determine whether the application of a peripheral proprioceptive stimulus to the neuromuscular motor points of the quadriceps increases strength and neuromuscular activation during the squat movement in the lower limbs of healthy, untrained subjects.

Methods: The design of this study is a randomized crossover clinical trial. All participants (n=36) will randomly receive both the Active and Sham proprioceptive stimulation.The proprioceptive stimulus will consist of intermittent mechanical pressure on the skin, localized at the neuromuscular motor points of the rectus femoris, vastus lateralis, and vastus medialis of the quadriceps. The tissue subjected to precise pressure in these highly innervated neuromuscular zones promotes the stimulation of kinesthetic cortical sensitivity. The outcome variable will be the assessment of Maximum Strength (MS) generated by the participant during the squat movement, from a 90º knee flexion position to full extension. At the moment of peak force, the mean velocity (MV) of the concentric phase of the movement and the maximum load the participant can move will be evaluated. The intervention, assessment, and recruitment will take place at the Faculty of Health Sciences, Blanquerna - Ramon Llull University

ELIGIBILITY:
Inclusion criteria :

* State of health with no history of neuromuscular injuries
* Without surgical interventions, or lower limb trauma in the last six months
* No associated cardiovascular disease
* No associated severe COPD.
* AllParticipants are considered untrained if they do not engage in any specific vigorous lower-limb strength training or regularly perform physical exercise or sports activities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Strength (MS) | estimated time of movement and data collection of 20 minutes
  The outcome variable will consist of the assessment of Maximum Strength (MS) generated by the participant during the squat movement, from a 90º knee flexion position to full extension measured in two units, kilograms and newtons.

OTHER OUTCOMES:
electric neuromuscular activation | estimated time of movement and data collection of 20 minutes
  In addition to strength assessment, portable sensors will be placed to digitize kinematics (knee and foot joint angles) and muscle electrical activity (surface electromyography), related to the variable of neuromuscular activation during the squat movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Pedro Victor López Plaza, Barcelona, Spain